CLINICAL TRIAL: NCT03590795
Title: VISC-Q Trial (Validation of an Online Sleep Characterization Questionnaire)
Status: Completed | Type: Observational
Sponsor: Philips Respironics (Industry)
Collaborators: Cooperative Research Center (CRC) for Alertness, Safety and Productivity (Unknown)
Responsible Party: Sponsor
Other Study IDs: SRC-AI-SC-2018-10138
Record Dates: First submitted 2018-07-10; First posted 2018-07-18 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Sleep

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Problem Sleepers: Those individuals that have self identified as having a unspecified sleep problem will take the sleep survey.
  Interventions: Other: Sleep survey

INTERVENTIONS:
Other: Sleep survey — The Sleep survey was created by the Collaborative Research Center (CRC), a joint effort of the Australian Government, Academia and Industry [including Philips]).

SUMMARY:
Sleep is an important contributing factor to people's health. However, over one third of the general population has sleep complaints, causing both health related problems, and economic impact. Many do not think their problem sleep is serious enough to consult a physician (primary care or sleep specialist). For a selection of this population, self-tracking devices can be a solution, but these trackers are often activity based and therefore lacking in their capacity to give insight into underlying causes of poor quality sleep and daytime fatigue.

A new options for these confused sleeper is an online questionnaire, developed by Philips and Cooperative Research Center (CRC) for Alertness, Safety and Productivity Imagine a troubled sleeper awake at 3 am, they search "Why can't I sleep?" and find the survey. From there the user takes the sleep survey, which has the ability to assess their most likely sleep problem or problems from a list of seven sleep problem categories based upon their responses. At the end of the survey, participants will get information about which problem category they will fall into, and the level of certainty around that.

The purpose of the study is to determine the accuracy of the questionnaire in identifying the correct sleep problem when compared with the assessment of a sleep physician in a clinical sleep center. We hope to enroll 200 participants which was based upon an Initial power analyses were completed using pilot data, assuming accuracy rates of 70, 80, and 90% and a total sample size of 200. The intervals would be about ± 4.5% (for 90%) to ± 7% (for 70%). Participants will complete the survey, be blinded to the results, and then have a consultation with a sleep physician who will make an independent assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age: 20-75 years old.
* Able to provide written informed consent
* Able to read, write and speak English

Exclusion Criteria:

* Has seen a sleep physician previously for formal clinical evaluation of a potential sleep problem.
* Is being treated for any sleep disorder.
* Has a major psychiatric disorder that is unstable at the time of evaluation.
* Has a major medical condition likely to contribute to and thus to confound any sleep problem (congestive heart failure, severe Chronic Obstructive Pulmonary Disease (COPD), a pain syndrome, etc).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be those who are new patients to the sleep lab or those recruited from a central recruiter that may or may not have sleep issues.
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2018-06-19 (Actual); Primary Completion 2018-09-07 (Actual); Study Completion 2018-09-07 (Actual)

PRIMARY OUTCOMES:
The primary analysis will calculate the agreement between the physician's primary diagnosis (considered the gold standard) and the Sleep survey's primary classification | 1 day
  The primary analysis will calculate the agreement between the physician's primary diagnosis (considered the gold standard) and the Sleep survey's primary classification. Percent agreement will be calculated for each sleep problem, and for the study sample as a whole, including the 95% confidence interval (CI).

SECONDARY OUTCOMES:
Percent agreement will be calculated to determine how often the survey includes the physician's primary diagnosis as one of its classifications. | 1 day
  Percent agreement will be calculated to determine how often the survey includes the physician's primary diagnosis as one of its classifications. This will be calculated for each sleep problem, and for the study sample as a whole, including the 95% confidence interval.

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Florida Lung & Sleep Associates, Lehigh Acres, Florida
  - NeuroTrials Research Inc., Atlanta, Georgia
  - Center for Sleep and Wake Disorders, Chevy Chase, Maryland
  - Clayton Sleep Institute, St Louis, Missouri
  - Sleep Therapy and Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
De-identified data sets will be shared with academic institutions for development purposes
Time Frame: After final study analysis data will be available for up to 5 years.